CLINICAL TRIAL: NCT01648049
Title: Treatment of Insomnia and Depression in Elders (TIDE)
Acronym: TIDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-0309; 1R34MH086643-01A2 (NIH)
Record Dates: First submitted 2012-06-26; First posted 2012-07-24 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Depression; Insomnia
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT (Experimental): Cognitive behavior therapy for both insomnia and depression featuring stimulus control and cognitive therapy.
  Interventions: Behavioral: Integrated Cognitive Behavioral Therapy (CBT)
- Treatment as Usual (Active Comparator): No additional treatment besides regular care.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Integrated Cognitive Behavioral Therapy (CBT) — CBT treatment is an abbreviated protocol based on manualized, evidence-based treatments for geriatric insomnia (Lichstein & Morin, 2000) and geriatric depression (Thompson, Gallagher-Thompson, & Dick, 1995).
  Arms: CBT
Behavioral: Treatment as usual — Standard Care - Treatment as usual
  Arms: Treatment as Usual

SUMMARY:
Insomnia and depression are two of the most prevalent mental health disorders and often co-occur.

Health disparities in rural America and among African-Americans are well documented. The investigators propose an R34 exploratory project to test the feasibility of delivering high-fidelity insomnia and depression psychological services to an underserved population. Treatment of Insomnia and Depression in Elders (TIDE) is a pilot study that will treat rural, predominantly African-American older adults who present to their primary care physician with co-occurring insomnia/depression. Stage 1 will be an uncontrolled case study series (n = 10) focusing on treatment development/refinement and patient acceptability. In stage 2, feasibility will be experimentally tested with 46 participants randomized to integrated cognitive-behavior therapy (CBT) + usual care or to usual care only in an effectiveness pilot study. The treatment will combine/integrate compact CBT for insomnia (including relaxation, sleep restriction, and stimulus control) and for depression (including cognitive therapy and behavioral activation). The experimental intervention comprises delivering CBT services by videoconferencing to patients in primary care settings who live in rural areas. Treatment will be evaluated by pre, post, and follow-up self report instruments on insomnia, depression, and quality of life. In addition, the stage 1 pilot will use investigator designed quantitative and qualitative measures to evaluate critical process variables including patient acceptability of the video format, patient acceptability of the treatments, and obstacles to adherence. Depending on stage 1 data, these measures may be incorporated into stage 2 as well. Several innovative features of this exploratory project include: intervening with CBT on both disorders hoping to gain a synergy by their combined presentation; use of telehealth to deliver treatment to distant locations; translation of efficacy findings to an effectiveness trial; treatment will be delivered in the primary care setting, the preferred locale of rural, older adults; the study will extend knowledge of the range of CBT applications by enrolling under-represented groups with respect to ethnicity, literacy, and financial resources.

The primary aims of this project are (1) to determine the feasibility and maximal therapy characteristics of integrated CBT for co-occurring insomnia/depression in both the case study series (stage 1) and the experimental investigation (stage 2), (2) collect pilot data on whether participants receiving integrated CBT + usual care show comparable or greater reductions in insomnia symptoms compared to participants receiving usual care at posttreatment and follow-up, and (3) collect pilot data on whether participants receiving integrated CBT + usual care show comparable or greater reductions in depression symptoms compared to participants receiving usual care at posttreatment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older,
* resident of the Black Belt or adjacent counties and receiving services from one of our primary care collaborators
* absence of significant cognitive impairment as indicated by a score of 24 or higher (17 or higher for those with only an eighth grade education) on the Mini-Mental Status Examination (MMSE; Folstein, Folstein, & McHugh, 1975
* not currently receiving psychological treatment,
* absence of serious suicidality
* concurrent psychiatric/medical disorders are not automatic disqualifiers unless they prevent participants from attending CBT therapy sessions or impede data collection,
* a referral from their primary care physician indicating presence of both insomnia and depression symptoms of sufficient significance to warrant initiation or continuance of primary care treatment for newly emergent or residual symptoms. Persons who are currently receiving pharmacotherapy for insomnia and/or depression must evidence residual symptoms of both disorders of sufficient magnitude to be evaluated as clinically significant and warranting further treatment by their primary care physician.

Exclusion Criteria:

* age is below 50
* not receiving services from one of our primary care collaborators
* significant cognitive impairment is present as indicated by a score of 23 or lower (16 or lower for those with only an eighth grade education) on the MMSE
* currently receiving psychological treatment
* presence of serious suicidality
* intrusive and unstable concurrent psychiatric/medical disorders
* primary care physician declines to refer

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | 3-month follow-up (23weeks post-treatment)
  Insomnia Measure
Hamilton Depression Scale | 10 weeks Post-treatment
  Depression measure
Hamilton Depression Scale | 3 Month follow-up (23 weeks post treatment)
  Depression Measure
Insomnia Severity Index | 10 weeks Post-treatment
  Insomnia Measure

SECONDARY OUTCOMES:
GDS | Pre-Treatment (Baseline/Week 0)
  Self-reported Geriatric Depression Scale
SOL | Pre-Treatment (Baseline/Week 0)
  self-reported Sleep Onset Latency
WASO | Pre-Treatment (Baseline/Week 0)
  Wake-time After Sleep Onset
SOL | 10 weeks Post-treatment
  Self-reported Sleep onset latency
SOL | 3-month follow-up (23weeks post-treatment)
  Self-reported Sleep onset latency
GDS | 10 weeks Post-treatment
  Self Reported Geriatric Depression Scale
GDS | 3-month follow-up (23weeks post-treatment)
  Self-reported Geriatric Depression Scale
WASO | 10 weeks Post-treatment
  Wake-time After Sleep Onset
WASO | 3-month follow-up (23weeks post-treatment)
  Wake-time After Sleep Onset

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L. Lichstein, Ph.D., Principal Investigator — University of Alabama, Tuscaloosa; Forrest Scogin, Ph.D., Principal Investigator — University of Alabama, Tuscaloosa
Locations (1):
- UATuscaloosa, Tuscaloosa, Alabama, United States